CLINICAL TRIAL: NCT01230671
Title: The Physical and Psychological Benefits of Yoga in Patients With Breast Cancer: A Feasibility Study
Brief Title: The Physical and Psychological Benefits of Yoga and Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Sarkis Meterissian (Other)
Responsible Party: Sponsor-Investigator, Dr. Sarkis Meterissian, Associate Dean, Faculty of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10-059-PSY
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): Patients in this arm will receive yoga therapy
  Interventions: Other: Yoga
- No yoga (Placebo Comparator): Patients will not have yoga in this arm

INTERVENTIONS:
Other: Yoga — A 12 week yoga session will be offered to women with breast cancer.
  Arms: Yoga

SUMMARY:
Breast Cancer is the most common cancer amongst Canadian women. Studies report that breast cancer patients are the most likely to use complementary medicine within the oncologic population. Yoga has become especially popular with this group as it promises to improve the mind, body and soul holistically. The investigators yoga program specifically focuses on rebuilding physical strength, increasing flexibility and reducing the pain and stress associated with the post-operative period. This study will examine how yoga can help improve the overall quality of life and its effects on the physical well-being of women with breast cancer. With positive statistical results, the investigators hope to implement yoga as part of their rehabilitation services at the Cedars Breast Clinic.

DETAILED DESCRIPTION:
Proposed Intervention:

1-hour hatha yoga classes, once a week for a 12-week period. One class will be offered in French, another in English. The class will begin with approximately 10 minutes of pranayama (breathing exercises) and meditation, followed by 30 minutes of yoga poses and ending with 10 minutes of sivasana (rest period.) The first couple of classes in the 12 week series will begin with restorative postures and will gradually progress to more gentle exercises. If health permits, the last couple of classes will involve some strengthening poses. A small portion of the class will work with the physical body in general and there will be a specific emphasis on the physical difficulties faced by most breast cancer patients, i.e. neck, chest, shoulders arms and hands.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-70
* Stage I to II breast cancer
* Minimum of 6 weeks Post Operative status

Exclusion Criteria:

* Previous/Current psychiatric history
* Concurrently involved in a yoga program
* Inability to undergo yoga training secondary to physical/health limitations outlined by the treating team

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Range of motion of the shoulders | 12 weeks
  The range of motion of the shoulders will be measured before and after the 12 week session and then compared.

SECONDARY OUTCOMES:
Anxiety | 12 weeks
  The participants will fill in questionnaires (HADS and the Distress Thermometer) before and after the 12 week session and the results will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedar's Breast Clinic, Royal Victoria Hospital, Montreal, Quebec, Canada